CLINICAL TRIAL: NCT05254080
Title: Assessing the Physiologic Effect of taVNS During a Cold Pressor Test
Brief Title: taVNS Cold Pressor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Christopher Austelle, Principal Investigator, Medical University of South Carolina
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 00113453; 5R25DA020537-15 (NIH)
Record Dates: First submitted 2022-01-18; First posted 2022-02-24 (Actual); Results first posted 2023-09-08 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: taVNS; Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active taVNS then Sham taVNS (Experimental): Participants will receive active then sham (placebo) ear stimulation.
  Interventions: Device: Active taVNS; Device: Sham taVNS
- Sham taVNS then Active taVNS (Experimental): Participants will receive sham (placebo) then active ear stimulation.
  Interventions: Device: Active taVNS; Device: Sham taVNS

INTERVENTIONS:
Device: Active taVNS — Electrodes will be attached to the participant's ear with a small sticker or clip, which will deliver mild stimulation. These electrodes will be plugged into the Digitimer DS7a device, which is a device that delivers transcutaneous auricular vagus nerve stimulation or taVNS. Stimulation will be delivered randomly to participant's tragus (the small cartilage knob before the ear canal) for up to 5 minutes while you participate in the stress induction test (by putting both feet into an ice bath).
Device: Sham taVNS — Electrodes will be attached to the participant's ear with a small sticker or clip, which will deliver mild stimulation. These electrodes will be plugged into the Digitimer DS7a device, which is a device that delivers transcutaneous auricular vagus nerve stimulation or taVNS. Stimulation will be delivered randomly to participant's tragus (the small cartilage knob before the ear canal) for up to 5 minutes while you participate in the stress induction test (by putting both feet into an ice bath). During sham (placebo) stimulation, ear electrodes will be attached to the participant's ear but they will not receive any stimulation.

SUMMARY:
This study explores the use of transcutaneous auricular vagus nerve stimulation (taVNS), a new form of neuromodulation which stimulates the ear. 24 healthy subjects without a past medical or psychiatric history will be recruited to participate in a phone screen followed by 1 lab visit. During the lab visit, subjects will participate twice in a validated stress induction technique called the cold pressor test, while concurrently receiving either active or sham taVNS. The cold pressor test consists of subjects placing their feet in an ice bath for a short period of time. Researchers will measure participant's heart rate while they receive taVNS (ear stimulation) and participate in the cold pressor test. Assessments of mood, anxiety, and stress will be collected at the beginning and end of the visit.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65 years
* English speaking
* Non-treatment-seeking community members

Exclusion Criteria:

* Diagnosis of COVID-19 in the past 14 days
* Facial or ear pain or recent ear trauma.
* Metal implant devices in the head, heart or neck.
* History of brain stimulation or other brain surgery.
* History of myocardial infarction or arrhythmia, bradycardia.
* Use of B-blockers, antiarrhythmic medication (sodium/potassium/calcium-channel blockers), or blood pressure medications.
* Active respiratory disorder.
* Personal or family history of seizure or epilepsy or personal use of medications that substantially reduce seizure threshold (e.g., olanzapine, chlorpromazine, lithium).
* Personal history of head injury, concussion, or self-report of moderate to severe traumatic brain injury.
* Individuals suffering from frequent/severe headaches.
* Individuals with a reported history of any mental health disorder or taking any psychotropic medications.
* Moderate to severe alcohol or substance use disorder.
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher W Austelle, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were excluded for any major medical comorbidities, as this study only enrolled healthy neurotypical participants. Upon enrollment, participants were automatically randomized to receive active taVNS or sham stimulation first (all participants received both active and sham, the order was randomized).
Period: Overall Study
Arm/Group | Active taVNS Then Sham taVNS | Sham taVNS Then Active taVNS
Started | 12 | 12
Completed | 10 | 11
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active taVNS Then Sham taVNS | Sham taVNS Then Active taVNS | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.75 (5.48) | 29 (5.24) | 28.38 (5.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Mean Heart Rate (Before CPT/taVNS)
Description: Heart rate will be measured with EKG electrodes before concurrent stress test and ear stimulation.
Time Frame: Baseline (up to 10 minutes prior to concurrent stress test and ear stimulation)
Measure: Mean (Standard Deviation); unit: beats per minute
Groups:
- Active taVNS: Participants will receive active ear stimulation.
  Active taVNS: Electrodes will be attached to the participant's ear with a small sticker or clip, which will deliver mild stimulation. These electrodes will be plugged into the Digitimer DS7a device, which is a device that delivers transcutaneous auricular vagus nerve stimulation or taVNS. Stimulation will be delivered randomly to participant's tragus (the small cartilage knob before the ear canal) for up to 5 minutes while you participate in the stress induction test (by putting both feet into an ice bath).
- Sham taVNS: Participants will receive sham (placebo) ear stimulation.
  Sham taVNS: Electrodes will be attached to the participant's ear with a small sticker or clip, which will deliver mild stimulation. These electrodes will be plugged into the Digitimer DS7a device, which is a device that delivers transcutaneous auricular vagus nerve stimulation or taVNS. Stimulation will be delivered randomly to participant's tragus (the small cartilage knob before the ear canal) for up to 5 minutes while you participate in the stress induction test (by putting both feet into an ice bath). During sham (placebo) stimulation, ear electrodes will be attached to the participant's ear but they will not receive any stimulation.
Arm/Group | Active taVNS | Sham taVNS
Number analyzed (Participants) | 21 | 21
beats per minute | 72.86 (10.88) | 72.0 (11.77)

2. Primary Outcome: Mean Heart Rate (During CPT/taVNS)
Description: Heart rate will be measured with EKG electrodes during concurrent stress test and ear stimulation.
Time Frame: During concurrent stress test and ear stimulation (average duration of 5 minutes)
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Active taVNS | Sham taVNS
Number analyzed (Participants) | 21 | 21
beats per minute | 83.54 (16.24) | 83.96 (16.35)

3. Primary Outcome: Mean Heart Rate (After CPT/taVNS)
Description: Heart rate will be measured with EKG electrodes after concurrent stress test and ear stimulation.
Time Frame: After concurrent stress test and ear stimulation (up to 10 minutes after concurrent stress test and ear stimulation)
Measure: Mean (Standard Deviation); unit: beats per minute
Groups:
- Sham taVNS: Participants will receive sham (placebo) stimulation.
  Sham taVNS: Electrodes will be attached to the participant's ear with a small sticker or clip, which will deliver mild stimulation. These electrodes will be plugged into the Digitimer DS7a device, which is a device that delivers transcutaneous auricular vagus nerve stimulation or taVNS. Stimulation will be delivered randomly to participant's tragus (the small cartilage knob before the ear canal) for up to 5 minutes while you participate in the stress induction test (by putting both feet into an ice bath). During sham (placebo) stimulation, ear electrodes will be attached to the participant's ear but they will not receive any stimulation.
Arm/Group | Active taVNS | Sham taVNS
Number analyzed (Participants) | 21 | 21
beats per minute | 68.97 (8.65) | 68.78 (9.54)

4. Secondary Outcome: Mean Score of Pain (Before CPT/taVNS)
Description: Pain will be assessed using a 0-10 scale (where 0 represents no pain at all and 10 represents the worst pain possible) before concurrent stress test and ear stimulation.
Time Frame: Baseline (up to 10 minutes prior to concurrent stress test and ear stimulation)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active taVNS | Sham taVNS
Number analyzed (Participants) | 21 | 21
units on a scale | 0.05 (0.22) | 0 (0)

5. Secondary Outcome: Mean Score of Pain (During CPT/taVNS)
Description: Pain will be assessed using a 0-10 scale (where 0 represents no pain at all and 10 represents the worst pain possible) during concurrent stress test and ear stimulation.
Time Frame: During concurrent stress test and ear stimulation (average duration of 5 minutes)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active taVNS | Sham taVNS
Number analyzed (Participants) | 21 | 21
units on a scale | 5.67 (2.39) | 5.62 (2.11)

6. Secondary Outcome: Mean Score of Pain (After CPT/taVNS)
Description: Pain will be assessed using a 0-10 scale (where 0 represents no pain at all and 10 represents the worst pain possible) after concurrent stress test and ear stimulation.
Time Frame: After concurrent stress test and ear stimulation (up to 10 minutes after concurrent stress test and ear stimulation)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active taVNS | Sham taVNS
Number analyzed (Participants) | 21 | 21
units on a scale | 0.24 (0.44) | 0.10 (0.30)

7. Secondary Outcome: Mean Score of Anxiety (Before CPT/taVNS)
Description: Anxiety will be assessed using a 0-10 scale (where 0 represents no anxiety at all and 10 represents the worst anxiety possible) before concurrent stress test and ear stimulation.
Time Frame: Baseline (up to 10 minutes prior to concurrent stress test and ear stimulation)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active taVNS | Sham taVNS
Number analyzed (Participants) | 21 | 21
units on a scale | 1.43 (1.72) | 1.81 (1.75)

8. Secondary Outcome: Mean Score of Anxiety (During CPT/taVNS)
Description: Anxiety will be assessed using a 0-10 scale (where 0 represents no anxiety at all and 10 represents the worst anxiety possible) during concurrent stress test and ear stimulation.
Time Frame: During concurrent stress test and ear stimulation (average duration of 5 minutes)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active taVNS | Sham taVNS
Number analyzed (Participants) | 21 | 21
units on a scale | 3.52 (2.77) | 3.48 (2.27)

9. Secondary Outcome: Mean Score of Anxiety (After CPT/taVNS)
Description: Anxiety will be assessed using a 0-10 scale (where 0 represents no anxiety at all and 10 represents the worst anxiety possible) after concurrent stress test and ear stimulation.
Time Frame: After concurrent stress test and ear stimulation (up to 10 minutes after concurrent stress test and ear stimulation)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active taVNS | Sham taVNS
Number analyzed (Participants) | 21 | 21
units on a scale | 0.48 (0.75) | 0.62 (0.92)

10. Secondary Outcome: Mean Score of Distress (Before CPT/taVNS)
Description: Distress will be assessed using a 0-10 scale (where 0 represents no distress at all and 10 represents the worst distress possible) before concurrent stress test and ear stimulation.
Time Frame: Baseline (up to 10 minutes prior to concurrent stress test and ear stimulation)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active taVNS | Sham taVNS
Number analyzed (Participants) | 21 | 21
units on a scale | 0.29 (1.10) | 0.33 (1.15)

11. Secondary Outcome: Mean Score of Distress (During CPT/taVNS)
Description: Distress will be assessed using a 0-10 scale (where 0 represents no distress at all and 10 represents the worst distress possible) during concurrent stress test and ear stimulation.
Time Frame: During concurrent stress test and ear stimulation (average duration of 5 minutes)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active taVNS | Sham taVNS
Number analyzed (Participants) | 21 | 21
units on a scale | 4.52 (3.04) | 4.48 (3.01)

12. Secondary Outcome: Mean Score of Distress (After CPT/taVNS)
Description: Distress will be assessed using a 0-10 scale (where 0 represents no distress at all and 10 represents the worst distress possible) after concurrent stress test and ear stimulation.
Time Frame: After concurrent stress test and ear stimulation (up to 10 minutes after concurrent stress test and ear stimulation)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active taVNS | Sham taVNS
Number analyzed (Participants) | 21 | 21
units on a scale | 0.05 (0.22) | 0.14 (0.36)

ADVERSE EVENTS:
Time Frame: 2 hours
Arm/Group | Active taVNS | Sham taVNS
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/80/NCT05254080/Prot_001.pdf
  • Informed Consent Form (2022-08-12): https://cdn.clinicaltrials.gov/large-docs/80/NCT05254080/ICF_002.pdf